CLINICAL TRIAL: NCT00237055
Title: Infectious Agents in Pediatric Crohn's Disease
Brief Title: Infectious Agents in Pediatric Crohn's
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: R03 DK64544 (completed); NIDDK R03 DK64544; R03DK064544 (NIH)
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
Keywords: Children; Crohn's disease; Inflammatory bowel disease; Infectious agents; Colonoscopy
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Six sites of the Pediatric Inflammatory Bowel Disease Consortium (plus 2 additional sites) will participate in this study. The participating sites will be that of the Principal Investigator (PI), Emory University School of Medicine, Atlanta, GA (Benjamin D. Gold, MD); Texas Children's Hospital / Baylor College of Medicine (George Ferry, MD and Tony Olive, MD); Children's Hospital of Philadelphia, Philadelphia, PA (Bob Baldassano, MD); University of Chicago Children's Hospital, Chicago, IL (Barbara Kirschner, MD); University of California, San Francisco (Mel Heyman, MD); Mass General Hospital / Harvard University (Harland Winter, MD); V.A. Stanford University School of Medicine, Stanford, CA (David Relman, MD); Children's Center For Digestive Healthcare, Atlanta, GA (Stanley Cohen, MD); and Centers for Disease Control and Prevention, Atlanta, GA (Drs. Jeannette Guarner, Siobhan O'Connor and Thomas Shinnick)

The duration of study is 2 yrs.

Objectives:

1. Improve the methods to collect biopsies from the colon and ileum, tissue storage techniques and best methods to detect specific infections in children with Crohn's disease;
2. Determine if there are specific infectious agents that are more common in children with Crohn's disease, and;
3. Determine if there are types of children with Crohn's disease (e.g., children living in Boston, African American children) who may be more at risk for getting the infections.

The study design involves children ages 6 months through 17 11/12 years of age who are undergoing a clinically-indicated colonoscopy. Subjects will be grouped into cases and controls.

* Any child ages 6 mos through 17 11/12 years of age, undergoing a clinically-indicated colonoscopy as determined by the treating physician, is eligible for enrollment. About 500 patients will be enrolled in this study.
* Cases will consist of those children within the defined age group, who are undergoing diagnostic colonoscopy and have the definitive diagnosis of Crohn's disease.
* Children who have the diagnosis of indeterminate colitis or ulcerative colitis for the purpose of this R03, will be excluded as cases and from initial analysis, but will have tissue specimens banked for subsequent evaluation for infectious agents.
* Controls will consists of children within the defined age group, undergoing clinically indicated colonoscopy and who are not diagnosed with Crohn's disease, ulcerative colitis or indeterminate colitis (e.g., juvenile polyps, irritable bowel syndrome or functional bowel disease).
* Stool specimen (5ml/1 tsp) will be collected to test for different types of bacteria
* A questionnaire will be administered to each research volunteer.
* Each subject's medical information (i.e. diagnosis, disease stage, and laboratory results) will be stored electronically in a separate access-based database. A unique identifier will be assigned to each patient entered into the study and will also be used for blinding of the specimens analyzed by the pathologist and by molecular assays for infectious agents.
* Colonoscopy will be performed by the treating pediatric gastroenterologist and biopsies obtained in the usual standard of care.
* Clinical biopsies from the rectum, left, right, transverse colon and cecum will be placed in formalin containing vials as per standard of care for the clinical pathologist and diagnostic evaluation.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), which includes CD and ulcerative colitis (UC), is estimated to affect approximately 1 - 2 million Americans. Recent studies strongly suggest that these disorders are increasing in prevalence in developed and developing countries, and in first generation immigrants to industrialized nations. Changing epidemiology of IBD implies that, in addition to a genetic susceptibility for disease, an environmental trigger or exposure likely impacts disease expression. However, the specific pathobiology and etiology of IBD remain unclear. Knowledge of the host genetic basis of IBD has advanced, including characterization of a novel susceptibility gene in adult and adolescent CD (NOD2/CARD-15) located on the pericentromeric region of chromosome 16. Recent studies not only implicate NOD2/CARD-15 in susceptibility to CD, but also suggest a link between the innate immune response to bacterial components and development of disease. Thus, well-designed investigations of infectious etiologies of CD, with sufficient power to detect differences in infection between IBD and non-IBD patients, are critically needed. Yet, deficiencies in the methods and tools for such studies still exist.

Both infectious and noninfectious mechanisms of pathogenesis remain plausible but unconfirmed. To date, scientific evidence cannot conclude whether one or more infectious pathogens triggers or determines the development and outcomes of CD or UC. Persistent exposure to "normal resident flora" in an abnormally permeable gut might also conceivably determine disease. Thus carefully designed investigations that apply systematically evaluated, reliable and reproducible detection assays are needed to confirm or disprove infectious hypotheses of causation. The first step is a pilot study that validates study design and complementary assays (morphology-, molecular- and culture-based) and uniformly applies these to target patient and control tissues (i.e., pediatric endoscopic biopsies). It must focus on newly diagnosed CD (surrogate for "incident" CD) in a well-characterized group of patients and appropriate, well-selected controls who meet uniform case and control definitions. It must develop reproducible methods to ensure that results from different studies can be compared and appropriate clinical interpretations made in order to translate research results into treatment and prevention strategies that decrease the burden of CD. At this time, deficiencies in both methodology and laboratory technology impede successful conduct and interpretation of the needed studies on causality.

Based on age of onset, newly diagnosed children with IBD, may be closer to triggering immunopathogenic events that initiate the inflammatory response than adults. They may also represent a unique population for the study of environmental factors (e.g., infection), i.e., younger age usually brings shorter and less complicated exposure histories to confound analyses. It is reasonable to postulate that a single agent or polymicrobial insults, in the genetically susceptible host, may determine the development or course of CD and it may be easier to identify some infectious determinants in childhood CD. We hypothesize that adequate collection of intestinal tissue biopsies from uniformly defined pediatric CD cases and controls and validation of sensitive and specific laboratory tools to detect potential infectious triggers of CD in these particular specimen types are needed to test causality for infection in CD. The Pedi IBDC, 6 large, geographically diverse U.S. centers represents an excellent platform to investigate potential infectious factors in CD, annually evaluating and recording clinical and epidemiologic data on ~288 newly diagnosed pediatric CD cases in a comprehensive data repository. The Pedi IBDC has a system to assess the safety and efficacy of its research. The Consortium also provides a pool of cases and controls in which to implement standardized specimen collection techniques under a well-conceived algorithm. The R03 assembled research team draws on a wide range of expertise and institutional resources in epidemiology, infectious disease pathology, molecular microbiology, mycobacteriology and virology, and the conduct of clinical trials. The multi-disciplinary expertise of this proposal can test and validate in small endoscopic biopsies the histopathology and molecular microbial detection assays previously validated in alternative paraffin-embedded or frozen tissues.

The R03 funding mechanism will facilitate tissue collection and banking techniques and evaluations of a panel of assays to detect select infectious agents ranging from those thought not to cause CD to those speculated as etiologic, from non-pathogenic commensals to known and undetermined pathogens. Therefore, our specific study aims are to:

1. standardize the collection (e.g., anatomic site of biopsy origin, biopsy number and collection technique), processing and banking of gastrointestinal tissue biopsies obtained during clinically-indicated endoscopy of well-characterized children with CD followed by the Pedi IBDC;
2. verify and standardize the definition of appropriate controls, evaluating both "non-diseased" biopsies from cases and clinically-indicated biopsies from children without IBD (e.g., juvenile polyposis, Hirschsprung's disease) to improve the design of future studies;
3. standardize and validate in pediatric biopsies detection methods to identify potential infectious risk factors for CD through parallel, paired and complementary pathology-based (IHC), broad range amplification-based molecular (PCR) and organism-specific (e.g., MAP) molecular analysis, and primary culture of tissue specimens taken from well-defined cases and controls.

Additionally, molecular characterization of microbiota in the feces from cases and controls will be compared to microbial detection in their respective tissue biopsies. Successful completion of these goals will provide a platform for imminent comprehensive investigations that characterize clinically relevant microbial risk factors for CD in the child and quite possibly the adult patient.

ELIGIBILITY:
Inclusion Criteria:

Each subject must satisfy all of the following inclusion criteria to be considered eligible for entry into this study:

1. Patients may be male or female 6 months though 17 11/12 years of age.
2. Patients must be undergoing clinically indicated colonoscopy at the discretion of their treating pediatric gastroenterologist.
3. Subject's parent or guardian must provide written informed consent, and children who are deemed old enough by the PI at each site must provide informed assent.

Exclusion Criteria:

Patients with any of the following characteristics will NOT be eligible for entry into the study:

1. Children who are determined to have the diagnosis of indeterminate colitis or ulcerative colitis for the purpose of this R03 - 2-year study will be excluded as cases and from the initial analysis, but will have tissue specimens banked for subsequent evaluation for infectious agents.
2. Patient has parent or guardian who refuses to sign the consent form or is not able to give fully informed consent due to mental deficiency or language problems.
3. Child who is deemed old enough to give assent and refuses to participate.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2004-08; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D. Gold, M.D., Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine; Emory Children's Center, Atlanta, Georgia, United States